CLINICAL TRIAL: NCT01119196
Title: The Measurement of Insulin Resistance in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100177
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal Dialysis; Insulin resistance
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glucose-based dialysate (No Intervention): most frequently used Standard of Care (SOC) dialysate
- Icodextrin dialysate (Other): alternate SOC dialysate
  Interventions: Other: Icodextrin dialysate

INTERVENTIONS:
Other: Icodextrin dialysate — use of alternate SOC dialysate
  Arms: Icodextrin dialysate

SUMMARY:
The goal of this study is to examine the relevance of insulin resistance in peritoneal dialysis (PD) patients as well as the means to improve this metabolic derangement. We will do so through a prospective randomized study using Icodextrin as an alternate dialysate solution to routine glucose-based dialysate. We hypothesize that (1) the glucose loading associated with PD leads to impairment in insulin sensitivity, (2) the degree of insulin resistance is dependent on the basal metabolic state (fasting versus stimulated), and (3) the replacement of conventional dialysate with glucose-sparing dialysate preparations will improve insulin resistance and associated metabolic disturbances in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and receiving stable PD for ≥ 3 months;
* BMI ≤ 45;
* Most recent Kt/V ≥1.7 or Tccr ≥ 50l/week/1.73m2;
* On Glucose lactate-buffered PD solutions with consistent glucose exposure.

Exclusion Criteria:

* Pregnancy or breast-feeding;
* Intolerance to the study protocols;
* Severe, unstable, active, or chronic inflammation disease (active infection, active connective tissue disorder, active cancer, HIV, liver disease);
* Chronic use of anti-inflammatory medication except low dose (< 10mg/d) prednisone;
* Severe hypokalemia (K+ level < 3.0 mEq/L);
* Hypercalcemia (Ca++ level > 11.0 mg/dL);
* Have a glycogen storage disease;
* Intolerant to maltose or isomaltose;
* Allergic to cornstarch or icodextrin;
* Recent abdominal surgery in the past 30 days;
* Chronic Obstructive Lung Disease (COPD) or Interstitial lung disease;
* Insulin-Dependent Diabetes Mellitus (IDDM).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
improvement in glucose disposal rate | 12 weeks

SECONDARY OUTCOMES:
the Pearson or Spearman correlation coefficient values between insulin resistance (IR) measured by insulin clamp study and other methods (e.g., HOMA, QUICKI, OGTT) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States